CLINICAL TRIAL: NCT06193694
Title: Coaching Program to Address Burnout, Wellness and Professional Development in Early Career Pediatric Surgeons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Healthcare System (Other)
Collaborators: Vanderbilt University Medical Center (Other); Harvard Medical School (HMS and HSDM) (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Coaching RCT
Record Dates: First submitted 2023-12-08; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Well-Being, Psychological; Surgical Residents; Burnout, Professional
MeSH Terms: conditions — Psychological Well-Being; Burnout, Professional

STUDY DESIGN:
Intervention Model Description: Early career pediatric surgeons will be randomized, in a 1:1 fashion to either receive wellness materials or formal coaching as described above.
  Randomization will occur after coaches are identified and have completed training in a 2:1 fashion to either participate as coaches or receive wellness materials.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive wellness materials (No Intervention): Control group - 50% of the study early career pediatric surgeon population will be randomized to the control group in a 1:1 manner after baseline burnout data is obtained. 33% of the coaches who volunteer will also be randomized to a control group in a 1:2 manner after baseline burnout data is obtained.
- Formal Coaching (Experimental): Study group - 50% of the study population will be randomized to the intervention or coaching group in a 1:1 manner after baseline burnout data is obtained. Similarly, 67% of the coaches who volunteer will be randomized to the intervention or coaching group in a 2:1 manner after baseline burnout data is obtained.
  Interventions: Behavioral: Coaching

INTERVENTIONS:
Behavioral: Coaching — Formal coaching program followed by the Coaching Fidelity Tool, to be taken by the study group after program completion contains 12 questions, predominantly multiple choice and yes/no, although there is one question that requires a short answer as well as a place to write additional comments. These questions are meant to elicit responses about their experience with their assigned coach during their one-on-one coaching sessions.
  Arms: Formal Coaching

SUMMARY:
Coaching is a useful tool that uses positivity and goal directed behaviors to increase resiliency and reduce physician burnout.

Objectives: Based on the principles of positive psychology, the objectives of the study are to improve early career pediatric surgeon (as defined by years 1-3 out of training) well- being, workplace satisfaction, decrease burnout and improve resiliency of both the coaches and early career pediatric surgeons.

DETAILED DESCRIPTION:
Coaching is used in business and many other career paths to help the individual define and create their own goals and strategies for achieving those goals. The Professional Development Coaching Program applies this model to help our residents in their professional development as physicians. While early career pediatric surgeons may have multiple evaluators and mentors, a coaching program provides them the opportunity for a nonsupervisory American Pediatric Surgical Association member to assist them in purely a coaching role. This program is based on the Massachusetts General Hospital Coaching program that was successfully developed and rolled out in 2011. This program was evaluated from 2012-present, and based on its success, it has since been adopted by >20 internal medicine residency programs around the country. Additionally, a similar program was piloted in 2018 to evaluate the program's success with remote coaching through the Association of Women Surgeons and the investigators have completed a program with remote coaching of pediatric surgery trainees by American Pediatric Surgical Association members that is now ongoing as a quality review project. The investigators would like to pursue a randomized coaching intervention and evaluation across early career pediatric surgeons to understand the impact of this program and its generalizability to surgical subspecialties and surgeons in the first 3 years of practice.

The goal of the Professional Development Coaching Program is to allow early career pediatric surgeons to understand their development over time, find meaning and purpose in their work, and identify their strengths and how to use these to overcome challenges and stressors. Additionally, the program connects early career pediatric surgeons with a seasoned faculty member who will work with them, grow to know them in-depth over time, and provide meaningful guidance throughout the relationship. There is an additional benefit to the coaches themselves, who are able to connect with other faculty coaches in a rewarding way that provides faculty development in leadership development and positive psychology, and space to interact with a group of like-minded physicians.

The program design will be mirrored on the American Pediatric Surgical Association Trainee Coaching Program - Each early career pediatric surgeon is assigned a Professional Development Coach, who is an American Pediatric Surgical Association member from a different program than theirs who has volunteered their time as a coach and has previously participated in the trainee program, thus allowing them to have more advanced coaching skills. Professional Development Coaches are assigned 1- 2 early career pediatric surgeons and are responsible for meeting with them quarterly to review evaluations, encourage reflection, provide guidance, and motivate them to set learning goals. Once early career pediatric surgeons are matched with their coach, they remain paired with their coach for the duration of the study (1 year). There is a one-year curriculum based on positive psychology and leadership development that is based on quarterly meetings. The faculty coaches receive 6 hours of training in positive psychology coaching during the study period.

Based on prior program evaluation, residents engage in the coaching program enthusiastically, and those who engage report lower levels of burnout, greater resiliency, greater satisfaction with their training experience, improved responses to stressors at work and in their personal life, and have increased opportunities for reflection and feedback. The investigators would like to study the Professional Development Coaching Program in this specific specialty and stage of practice, as it differs from prior evaluations, by engaging in a randomized trial comparing coaching to usual mentoring and well-being practices, and if successful, provide an opportunity for crossover in year 2 where coaching is then extended to all early career pediatric surgeons. This is unique in that coaching of peers can be challenging for novice coaches, thus this study seeks to study early career pediatric surgeons coached by coaches 6 or more years out of training who have had some prior coaching experience to see if this model is effective.

This study would be carried out through the American Pediatric Surgical Association network. All early career pediatric surgeons will be offered enrollment in the study. A baseline survey will be obtained to allow for randomization to either coaching, or usual mentoring and well-being practices that exist in the residency and/or fellowship. The investigators will quantitatively survey the early career pediatric surgeons and coaches regarding their experiences with and assessment of the Professional Development Coaching Program at the end of each year of the study period.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria for coaches include:

1. APSA members in good standing 6 or more years out of training who have participated in coaching through the APSA Trainee coaching project with interest in coaching who attend full online or in person training session in May of 2022.

Inclusion criteria for early career pediatric surgeons include:

1. North American early career pediatric surgeons who are interested in receiving coaching.

-

Exclusion Criteria: None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Examine the Impact of the Coaching Relationship in early career Pediatric Surgeons on well-being and burnout compared to non-coached controls. | 1 year
  All participants were asked to complete pre/post surveys using elements from validated measures: PERMA-profiler (5-pt Likert, {1-5}, 14 items, range 14-70. Score: Average of items comprising each; Professional Fulfillment Index (professional fulfillment in physicians, 5-point Likert {0-4}, 6 items, range 0-4) Burnout (5-point Likert {0-4}, 10 items, range 0-4); Scoring: Average of all items within each scale; Self-Valuation Scale (Prioritization: Personal well-being/ability to adopt a growth mindset, 5-point Likert {0-4}, 4 items, range 0-16); Gratitude Scale (7-point Likert {1-7}, 2 items, range 2-14); Intolerance of Uncertainty Scale emotional/cognitive/behavioral reactions to ambiguous situations; 5-point Likert {1-5}, 12 items, range 12-60); Dispositional Resilience Scale (hardiness, 4-point Likert {0-3}, 15 items, range 0-45), score: Sum of respective items; Measure of Current Status (Ability to deal with stress, 5-point Likert {0-4}, 3 items, range 0-12).

SECONDARY OUTCOMES:
Impact of Coaching on professional fulfillment | 1 year
  Examine the impact of the coaching relationship on early career pediatric surgeon's professional fulfillment, compared to non-coached controls - scales used as above for outcome #1
Effectiveness of coaching relationship among peers | 1 year
  Examine the effectiveness of a coaching relationship established among peers by employing a difference in career stage and repeated coach training - scales used as above for outcome #1
Effectiveness of coaching relationship on well-being and professional fulfillment | 1 year
  Examine the impact of the coaching relationship on coach well-being and professional fulfillment, compared to non-coach controls. Scales used as above for outcome #1.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Healthcare System, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data to be shared upon written request and at general American Pediatric Surgical Association meeting.